CLINICAL TRIAL: NCT07264738
Title: Oral Ondansetron to Improve Patient Experience of Unsedated Esophagogastroduodenoscopy: A Pilot Study
Brief Title: Oral Ondansetron to Improve Patient Experience of Unsedated Esophagogastroduodenoscopy Pilot Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Chief physician of Gastroenterology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ON-COMFORT25
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Esophagogastroduodensocopy (EGD) Procedure
MeSH Terms: interventions — Ondansetron; dyclonine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral ondansetron and dyclonine hydrochloride mucilage (Experimental)
  Interventions: Drug: ondansetron and dyclonine hydrochloride
- dyclonine hydrochloride mucilage only (Other)
  Interventions: Drug: dyclonine hydrochloride only

INTERVENTIONS:
Drug: ondansetron and dyclonine hydrochloride — Patients will take 8 mg oral ondansetron 2 hours prior to EGD process in addition to dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to EGD process.
  Arms: oral ondansetron and dyclonine hydrochloride mucilage
Drug: dyclonine hydrochloride only — Patients will be instructed to gurgle 10 mL of dyclonine chloride mucilage (0.01 g/mL) and gurgle for 1 minute 15 minutes prior to endoscopic process.
  Arms: dyclonine hydrochloride mucilage only

SUMMARY:
The goal of this interventional pilot study is to explore the feasibility of administering ondansetron prior to esophagogastroduodenoscopy (EGD), and preliminarily test if it can alleviate the gagging reflex, nausea and vomiting in Chinese patients undergoing unsedated diagnostic EGD. The main questions it aims to answer are:

Is adding oral ondansetron to pre-medication regimen of unsedated EGD safe, easy to conduct, and well-accepted by patients? May taking ondansetron prior to EGD reduce the discomfort of patients during the endoscopic process? May taking ondansetron prior to EGD reduce the intensity of patient gagging and nausea, and the incidence of vomiting ? Researchers will compare premedication of oral ondasetron and topical pharyngeal anesthesia (dyclonine hydrochloride mucilage) with topical pharyngeal anesthesia only to answer the questions above.

Participants will be treated with one of the following regimens according to the randomization result:

* Oral ondansetron of 8 mg 2 hours prior to endoscopic process and dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to endoscopic process;
* dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to endoscopic process.

After the endoscopic process is finished, patients will be asked to fill in a questionnaire that contains the following items, all measured by NRS 0-10:

* Overall discomfort;
* Intensity of gagging;
* Willingness to undergo unsedated EGD again if indicated.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for follow-up EGD at PUMCH
* Signing a written informed consent.

Exclusion Criteria:

* Contraindications for esophagogastroduodenoscopy.
* History of upper gastrointestinal tract surgery.
* With conditions indicated for emergency EGD, such as upper gastrointestinal bleeding
* Severe diseases of the heart, kidney, respiratory system, central nervous system, and hematopoietic system.
* Pregnancy.
* Neuropsychiatric disorders, severe depression and severe anxiety.
* Allergy to ondansetron or dyclonine hydrochloride.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in overall discomfort | from the previous endoscopy to 30 minutes after the current endoscopy is finished
  All 20 patients were follow-up patients who had unsedated EGD before. They assessed their degree of overall discomfort during the curent examination and the previous examination, both in NRS 0-10. Change in overall discomfort is the value of the difference between the previous and current NRS (previous-current).

SECONDARY OUTCOMES:
Change in patient gagging intensity | from the previous endoscopic examination to 30 minutes after the current examination is finished.
  Patients assessed their gagging intensity during the curent examination and the previous examination, both in NRS 0-10. Change in overall discomfort is the value of the difference between the previous and current NRS (previous-current).
Patient willingness to undergo unsedated EGD again | from start of endoscopy to 30 minutes after the examination is finished
  the willingness of patients to undergo unsedated EGD in the same method again, assessed by NRS 0-10 (0, not willing at all; 10 completely willing).
Intensity of patient gagging evaluated by endoscopist | from the start of the endoscopic process to the end of the endoscopic process
  measured by NRS 0-10, (0 none, 10 extremely strong) in a questionnaire given to endoscopists after the endoscopic process is finished
Endoscopist satisfaction for patient cooperation | from the start to the end of the endoscopic process
  satisfaction of endoscopist for patient cooperation in this process, assessed by NRS 0-10 (0, not satisfied at all; 10 very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No